CLINICAL TRIAL: NCT04232072
Title: Comparison of Intravenous Ibuprofen and Erector Spinae Plane Block for Postoperative Pain Management After Laparoscopic Sleeve Gastrectomy. A Randomized Controlled Study
Brief Title: Ibuprofen and Erector Spinae Plane Block After Laparoscopic Sleeve Gastrectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medipol Hospital 8
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Obesity
Keywords: Ibuprofen; Erector spina plane block; Postoperative analgesia management; Laparoscopic sleeve gastrectomy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: There are three models for this study. The first group is erector spinae plane block group, the second one is intravenous ibuprofen group, the third group is the no intervention control group
Who Masked: Outcomes Assessor
Masking Description: The anesthesiologist who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group ESPB = Erector spinae plane block group (Active Comparator): ESPB will be performed 30 min before induction of general anesthesia, with patients in the sitting position by using US. Under aseptic conditions, the high frequency linear probe will be covered with a sterile sheath and a 22G, 50 mm block needle will be used. Local anesthetic infiltration with 2% of lidocaine will be applied under the skin. US probe will be placed longitudinally 2-3 cm lateral to the T7 transvers process. The block needle will be inserted cranio caudal direction and then for correction of the needle 5 ml saline will be enjected deep into the erector spina muscle fascia. Following confirmation of the correct position of the needle 20 ml %0.25 bupivacaine will be administered for block. The same procedure will be performed for the opposite site.
  Interventions: Other: Group ESPB
- Group Ibuprofen = Ibuprofen (Active Comparator): In Group Ibuprofen, a dose of 800 mg ibuprofen IV will be administrated 30 min before induction of general anesthesia.
  Interventions: Other: Group Ibuprofen
- Group C = Control group (No Intervention): A dose of 100 mg tramadol intravenously will be performed to all patients 30 min before the end of the surgery for postoperative analgesia. At the end of the surgery, local anesthetic infiltration will be perfomed around the port entrance sites by the surgical team to the all patients. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit at the postoperative period.

INTERVENTIONS:
Other: Group ESPB — A dose of 100 mg tramadol intravenously will be performed to all patients 30 min before the end of the surgery for postoperative analgesia. At the end of the surgery, local anesthetic infiltration will be perfomed around the port entrance sites by the surgical team to the all patients. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit at the postoperative period.
  Arms: Group ESPB = Erector spinae plane block group
Other: Group Ibuprofen — A dose of 100 mg tramadol intravenously will be performed to all patients 30 min before the end of the surgery for postoperative analgesia. At the end of the surgery, local anesthetic infiltration will be perfomed around the port entrance sites by the surgical team to the all patients. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit at the postoperative period. In Group Ibuprofen, patients will be administered ibuprofen 800 mgr IV every 8 hours in the postoperative period.
  Arms: Group Ibuprofen = Ibuprofen

SUMMARY:
Laparoscopic sleeve gastrectomy (LSG) is defined as the first-step bariatric surgery for patients in the high surgical risk group. It has been shown that the laparoscopic approach has lower complication rates, shorter hospital stays, and earlier mobilization compared to open surgery. However, postoperative pain management is very important because it might cause major morbidity, especially pulmonary complications in the early postoperative period.

The intravenous (IV) form of ibuprofen has been used in the pain treatment since 2009. It has been shown to be effective, safe and with less adverse effects in the treatment of postoperative pain. It has been reported that ibuprofen provides effective postoperative pain management after LSG surgery.

The ultrasound (US) guided erector spina plane block (ESPB) is a novel interfacial plan block defined by Forero et al. ESPB provides thoracic analgesia at T5 level, abdominal analgesia at T7-9 level. In the literature, it has been reported that ESPB provides effective analgesia after LSG surgery.

The aim of this study is to compare US-guided ESPB and IV ibuprofen for postoperative analgesia management after LSG surgery.

DETAILED DESCRIPTION:
Bariatric surgery has been widely used in the treatment of obesity in recent years. Laparoscopic sleeve gastrectomy (LSG) is defined as the first-step bariatric surgery for patients in the high surgical risk group. It has been shown that the laparoscopic approach has lower complication rates, shorter hospital stays, and earlier mobilization compared to open surgery. However, postoperative pain management is very important because it might cause major morbidity, especially pulmonary complications in the early postoperative period. General recommendations for bariatric surgery include multimodal analgesia without sedatives, local analgesic infiltration, and early mobilization. Opioid analgesics are often preferred for pain management because of their strong analgesic potentials. However, opioids have undesirable adverse effects such as sedation, dizziness, constipation, nausea, vomiting, physical dependence and addiction, hyperalgesia, immunologic and hormonal dysfunction, muscle rigidity, tolerance, and respiratory depression. Therefore, the American Society of Anesthesiologists (ASA) recommends the use of multimodal analgesia including local anesthesia, regional anesthesia and nonsteroidal anti-inflammatory drugs (NSAIDs).

NSAIDs have long been used in the treatment of pain and inflammation. Ibuprofen is a propionic acid derivative that has anti-inflammatory, antipyretic, and analgesic effects similar to other NSAIDs. The intravenous (IV) form of ibuprofen has been used in the pain treatment since 2009. It has been shown to be effective, safe and with less adverse effects in the treatment of postoperative pain. It has been reported that ibuprofen provides effective postoperative pain management after LSG surgery.

The ultrasound (US) guided erector spina plane block (ESPB) is a novel interfacial plan block defined by Forero et al. The ESPB contains a local anesthetic injection into the deep fascia of erector spinae. This area is away from the pleural and neurological structures and thus minimizes the risk of complications due to injury. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. Cadaveric studies have shown that the injection spreads to the ventral and dorsal roots of the spinal nerves. ESPB provides thoracic analgesia at T5 level, abdominal analgesia at T7-9 level. In the literature, it has been reported that ESPB provides effective analgesia after LSG surgery.

The aim of this study is to compare US-guided ESPB and IV ibuprofen for postoperative analgesia management after LSG surgery. The primary aim is to compare postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for laparoscopic sleeve gastrectomy surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis,
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | Changes from baseline opioid consumption at postoperative 1, 2, 4, 8, 16 and 24 hours.
  The primary aim is to compare postoperative opioid consumption

SECONDARY OUTCOMES:
Pain scores (Visual analogue scores-VAS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16 and 24 hours.
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during mobilization will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Ciftci B, Ekinci M, Celik EC, Kaciroglu A, Karakaya MA, Demiraran Y, Ozdenkaya Y. Comparison of Intravenous Ibuprofen and Paracetamol for Postoperative Pain Management after Laparoscopic Sleeve Gastrectomy. A Randomized Controlled Study. Obes Surg. 2019 Mar;29(3):765-770. doi: 10.1007/s11695-018-3613-1. PMID 30474791
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016